CLINICAL TRIAL: NCT02273674
Title: Repetitive Transcranial Magnetic Stimulation in Borderline Personality Disorder Patients. Effects in Clinical Measurements, Inhibition, Cognitive Flexibility, and Social Cognition Process
Brief Title: TMS in Borderline Personality Disorder Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Psiquiatría Dr. Ramón de la Fuente (Other)
Collaborators: Universidad Nacional Autonoma de Mexico (Other)
Responsible Party: Principal Investigator, Julian Reyes Lopez, Medical doctor Psychiatry, Instituto Nacional de Psiquiatría Dr. Ramón de la Fuente
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SC-14-1006
Record Dates: First submitted 2014-10-15; First posted 2014-10-24 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Borderline Personality Disorder
Keywords: Borderline Personality Disorder; Transcranial Magnetic Stimulation, Repetitive
MeSH Terms: conditions — Borderline Personality Disorder

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Left rTMS 5 Hz (Experimental): This group receive transcranial magnetic stimulation at 5 Hz of frequency over left dorsolateral prefrontal cortex. Once a day on monday to friday. Until receive 15 sessions. After this the subjects, will be received 8 more sessions of TMS, one session at week for next eight weeks
  Interventions: Device: Left rTMS 5 Hz
- Right r TMS 1 Hz (Experimental): This group receive transcranial magnetic stimulation at 1 Hz of frequency over right dorsolateral prefrontal cortex. Once a day on monday to friday. Until receive 15 sessions. After this the subjects, will be received 8 more sessions of TMS, one session at week for next eight weeks
  Interventions: Device: Right r TMS 1 Hz

INTERVENTIONS:
Device: Left rTMS 5 Hz — The subjects will receive transcranial magnetic stimulation (5 Hz of frequency over left dorsolateral prefrontal cortex . Once a day on monday to friday. Until receive 15 sessions. After this the subjects, will be received 8 more sessions of TMS, one session at week for next eight weeks
  Arms: Left rTMS 5 Hz
Device: Right r TMS 1 Hz — The subjects will receive transcranial magnetic stimulation (1 Hz of frequency over right dorsolateral prefrontal cortex . Once a day on monday to friday. Until receive 15 sessions. After this the subjects, will be received 8 more sessions of TMS, one session at week for next eight weeks
  Arms: Right r TMS 1 Hz

SUMMARY:
The purpose of this study is to determine the potential effects of repetitive transcranial magnetic stimulation in the improvement of neuropsychological deficits and symptomatology in borderline personality disorder patients. Specially in cognitive flexibility, inhibition control and social cognition.

DETAILED DESCRIPTION:
This is a randomized, parallel group clinical trial to evaluate the efficacy of two protocols of repetitive Transcranial Magnetic Stimulation (rTMS), the application will be over dorsolateral prefrontal cortex (DLPFC) right and left, in patients with borderline personality disorder. 40 ambulatory patients with a borderline personality disorder diagnosis from the National Institute of Psychiatry in México will be included. All Patients will be randomly assigned and will complete a total of 23 sessions rTMS, in any of two groups:

5 Hz Group.- This group will receive rTMS sessions, 5 per week during three weeks (acute treatment phase), and after that, one session a week for the next eight weeks (follow up). The rTMS will be applied over the left DLPFC at 5 Hz, 1500 pulses per session in 100% of Motor threshold

1 Hz Group.- This group will receive rTMS sessions, 5 per week during three weeks (acute treatment phase), and after that, one session a week for the next eight weeks (follow up).

The rTMS will be applied over the right DLPFC at 1 Hz, 900 pulses per session in 100% of Motor threshold All sessions will be applied with a "Dantec" transcranial magnetic stimulator. The affective, borderline and anxiety symptoms will be evaluated at baseline, and every 5 TMS sessions during the acute treatment phase, and once at the end of the 8-weeks follow up. In same form for neuropsychological evaluations .

Categorical variables will be described by percentages and frequencies. Continuous variables will be described by means and standard deviations. Treatment groups will be compared using Student's T test. Cognitive, anxiety, borderline and affective symptom scale scores between treatment groups will be compared using repeated measures ANOVA

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of borderline personality disorder according to diagnostic and statistical manual of mental disorders IV text revision
* Treatment with selective inhibitors of serotonin reuptake
* Mass corporal index more than 19

Exclusion Criteria:

* Suicide risk or suicide attempt recent or actual
* History of epilepsy or seizures
* History of cranial trauma with loss awareness
* Intracranial or intraocular ferromagnetic devices, including skull prosthesis.
* Pregnant womens.
* Neurosurgery, cardiac pacemaker, lefthander
* Patients with psychotic symptoms, bipolar disorder or substance addiction.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2014-01; Primary Completion 2016-01 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in BORDERLINE EVALUATION OF SEVERITY OVER TIME (BEST) | Inclusion, after 15 days of treatment and at 8 weeks follow up
  The Borderline Evaluation of Severity Over Time (BEST) was developed to rate the thoughts, emotions, and behaviors typical of borderline personality disorder.

SECONDARY OUTCOMES:
Change from Baseline in Barratt impulsiveness scale | IInclusion, after 15 days of treatment and at 8 weeks follow up
  The Barratt Impulsiveness Scale is a questionnaire designed to assess the personality/behavioral construct of impulsiveness.
Change from Baseline in Hamilton Depression rating scale | Inclusion, after 15 days of treatment and at 8 weeks follow up
  The Hamilton depression rating scale is a is a multiple item questionnaire used to provide an indication of depression, and as a guide to evaluate recovery
Change from Baseline in Wisconsin card sorting test (WCST) | Inclusion, after 15 days of treatment and at 8 weeks follow up
  WCST is used primarily to assess perseveration and abstract thinking, the WCST is also considered a measure of executive function because of its reported sensitivity to frontal lobe dysfunction.
Change from Baseline in Stop Signal Task (SST) | Inclusion, after 15 days of treatment and at 8 weeks follow up
  SST measuring response inhibition (impulse control). The subject must respond to an arrow stimulus, by touching either of two choices depending on the direction in which the arrow points. If an audio tone is present, the subject must inhibit that response.
Change from Baseline in Reading the Mind in the Eyes Test | Inclusion, after 15 days of treatment and at 8 weeks follow up
  The 'Reading the Mind in the Eyes' (Eyes) test is an advanced test of theory of mind. It is widely used to assess individual differences in social cognition and emotion recognition across different groups and cultures.

CONTACTS AND LOCATIONS:
Overall Officials: Julian V Reyes, M.D., Principal Investigator — Instituto Nacional de Psiquiatria
Locations (1):
- Instituto Nacional de Psiquiatria Ramon de la Fuente, Mexico City, Mexico City, Mexico

REFERENCES:
- [Background] Arbabi M, Hafizi S, Ansari S, Oghabian MA, Hasani N. High frequency TMS for the management of Borderline Personality Disorder: a case report. Asian J Psychiatr. 2013 Dec;6(6):614-7. doi: 10.1016/j.ajp.2013.05.006. Epub 2013 Jun 14. PMID 24309885
- [Derived] Reyes-Lopez J, Ricardo-Garcell J, Armas-Castaneda G, Garcia-Anaya M, Arango-De Montis I, Gonzalez-Olvera JJ, Pellicer F. Clinical improvement in patients with borderline personality disorder after treatment with repetitive transcranial magnetic stimulation: preliminary results. Braz J Psychiatry. 2018 Jan-Mar;40(1):97-104. doi: 10.1590/1516-4446-2016-2112. Epub 2017 Jun 12. PMID 28614492